CLINICAL TRIAL: NCT00757354
Title: A Clinical Evaluation of Metal Ion Release From Metal-on-Metal Cementless Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Collaborators: Biomet U.K. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMETEU.CR.EU46
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Osteoarthritis; Avascular Necrosis; Traumatic Arthritis; Rheumatoid Arthritis
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis; Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metal on Metal cementless hip (Experimental): Metal on Metal cementless hip arthroplasty
  Interventions: Procedure: Metal on Metal cementless hip

INTERVENTIONS:
Procedure: Metal on Metal cementless hip — Metal on Metal hip arthroplasty
  Other Names: metal on metal hip arthroplasty

SUMMARY:
A clinical Evaluation to determine metal ion release from 4th generation metal-on-metal hip articulating surfaces in cementless total hip arthroplasty.

DETAILED DESCRIPTION:
This evaluation is being conducted to investigate the extent of metal ion release and its incorporation into the surrounding tissue resulting from metal on metal articulating surfaces in cementless total hip arthroplasty.

The amount of metallic ions released post operatively will be assessed by the concentration of Cobalt, Chromium and Molybdenum present in urine and analysed by I.C.P.M.S. (Inductive Coupled Plasma Mass Spectroscopy). The amounts of metallic ions released will be related to the hip function and range of motion measured pre-operatively and post-operatively. Secondary performance of the metal-on-metal articulation will be determined by radiographic evaluation and incidence of complications / revision rates.

ELIGIBILITY:
Inclusion Criteria:

* Subjects selected for this Evaluation will be grouped by initial diagnosis into one of the following diagnostic groups:

  * Non-inflammatory degenerative joint disease including osteoarthritis, avascular necrosis and traumatic arthritis.
  * Rheumatoid arthritis.
* Selection of subjects for this Evaluation should include the following considerations:

  * Patients under 70 years of age.
  * Willing to return for follow-up evaluations.
  * No bias to sex.

Exclusion Criteria:

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2012-06; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
concentration of Cobalt, Chromium and Molybdenum ions in urine | various follow-up visits

SECONDARY OUTCOMES:
harris Hip Score, oxford hip, WOMAC and SF-12 | various follow-up visits

CONTACTS AND LOCATIONS:
Overall Officials: Evert J Smith, FRCS, Principal Investigator — Avon Orthopaedic Centre
Locations (1):
- Avon Orthopaedic Centre, Bristol, United Kingdom